CLINICAL TRIAL: NCT05630157
Title: Evaluation of Effectiveness of the School-based Substance Use Prevention Program "Unplugged" on Gambling Behaviors Among Adolescents: an Experimental Controlled Study
Brief Title: Evaluation of Effectiveness of the Unplugged Program on Gambling Among Adolescents (GAPUnplugged)
Acronym: GAPUnplugged
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Università degli Studi del Piemonte Orientale Amedeo Avogadro (Other)
Collaborators: ASL Roma 1 (Unknown)
Responsible Party: Principal Investigator, Federica Vigna Taglianti, professor, Università degli Studi del Piemonte Orientale Amedeo Avogadro
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 080.742
Record Dates: First submitted 2022-11-17; First posted 2022-11-29 (Actual); Last update posted 2022-11-29 (Actual); Status verified 2022-11

CONDITIONS: Gambling
Keywords: Gambling; Prevention; School; Uplugged; Students; Effectiveness; Adolescents
MeSH Terms: conditions — Gambling

STUDY DESIGN:
Intervention Model Description: non randomized cluster controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Unplugged plus gambling component (Experimental): The experimental arm will receive the Unplugged curriculum plus a gambling component
  Interventions: Behavioral: Unplugged plus gambling component
- Usual curriculum (No Intervention): The Usual curriculum arm won't receive any specific prevention program

INTERVENTIONS:
Behavioral: Unplugged plus gambling component — 12 units/lessons of the Unplugged prevention curriculum plus a gambling component including specific gambling contents in units 3-4-5-7-9 and a 13th unit based on probability and mathematical concepts taught through an online simulator
  Other Names: GAPUnplugged
  Arms: Unplugged plus gambling component

SUMMARY:
The main aim of this study is to assess the effectiveness of a new component on gambling prevention to be added to the evidence-based school based prevention curriculum "Unplugged". The evaluation of effectiveness will be performed by conducting a non-randomized cluster controlled trial in classes of pupils 12 to 14 years old. Classes will be allocated to the intervention arm (receving Unplugged + the gambling component) or to the control arm (usual curriculum, no specific intervention).

The intervention includes 12 prevention units and a 13th unit focused on gambling. It will be carried out by Unplugged teachers trained in a specific training course. Data collection will take place before and after the intervention through a standardized questionnaire developed ad hoc and containing previously validated questions.

DETAILED DESCRIPTION:
The goals of the present non-randomized cluster controlled experimental trial (CCT) with follow-up at 4-8 weeks after the end of the intervention are:

1. to assess the effectiveness of a gambling-focused component added to the Unplugged prevention curriculum on: gambling behaviors, knowledge, attitudes, risk perceptions, beliefs, refusal skills, and normative perceptions;
2. to estimate the prevalence of gambling behaviors among Italian adolescents aged 12 to 14 years.

Unplugged is a school-based curriculum aimed to prevent tobacco, alcohol and drugs use among adolescents, developed and tested in the EUDap trial (www.eudap.net). It was demonstrated to be effective in several studies (Faggiano 2007; 2008; 2010; Gabrhelik 2012; Sanchez 2021; Vigna-Taglianti 2021) and included among evidence-based prevention programs (EMCDDA; Foxcroft 2011; Catalano 2012).

Secondary schools in Lazio, Piedmont and other Italian regions will be invited to take part in the study. Participation is voluntary for both the intervention and the control group. The schools participating in the study will inform caregivers and ask their consent for the participationof students and the data collection. Only students whose caregivers have given consent to participate will be involved in the study which will last about 7 months. The first questionnaire will be administered between November and December 2022 both in the control and the intervention group. Afterwards, the intervention group will received the 12 units of the Unplugged program and the gambling component, for about 3 months. Finally, after 4 to 8 weeks from the completion of the program, the same evaluation questionnaire will be administeres both in the control and in the intervention classes.

The questionnaire will be anonymous and will report only a pseudo-anonymization code for linkage of baseline and follow-up data. At the end of the survey, data will be analyzed in aggregated and anonymized form.

ELIGIBILITY:
Inclusion Criteria:

* Schools/classes in which at least one teacher has participated in the training course for Unplugged teachers, either in the past or in the weeks before the beginning of the study.
* Participation of already trained teachers in a booster training session on the gambling component.

Exclusion Criteria:

* classes which already started the Unplugged program in fall 2022, before the start of the study.
* pupils whose caregivers expressed refusal to participate in the study.

Ages: 12 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 3046 (Estimated)
Dates: Start 2022-11-21 (Estimated); Primary Completion 2023-11-21 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Prevalence of gambling behaviors | follow-up (4-8 weeks after completion of intervention)
  past 30 days frequency of gambling behaviors

SECONDARY OUTCOMES:
Prevalence of at-risk gambling behavior | follow-up (4-8 weeks after completion of intervention)
  past 30 days frequency of at risk indicator according to the definition of SOGS-RA (Wiebe 2000)
Beliefs about gambling | follow-up (4-8 weeks after completion of intervention)
  score of the 7 items scale assessing false beliefs concerning gambling (e.g. "If I gamble often, I have a greater chance of winning").
Attitudes towards gambling | follow-up (4-8 weeks after completion of intervention)
  score of the 6 items scale assessing attitudes about gambling by asking "What do you think about gambling" (e.g. "I think gambling is fun").
Refusal skills for gambling | follow-up (4-8 weeks after completion of intervention)
  proportion of pupils answering they will refuse vs accept the proposal of gambling from a friend (three scenarios)
Normative perceptions on gambling | follow-up (4-8 weeks after completion of intervention)
  proportion of pupils scoring as >50% the proportion of friends or people of their age who gamble
Risk perceptions on gambling | follow-up (4-8 weeks after completion of intervention)
  proportion of pupils with high vs low risk perceptions towards gambling as measured by a question asking "How much do you think people arm themselves by gambling to.."

CONTACTS AND LOCATIONS:
Overall Officials: Federica D Vigna-Taglianti, PhD, Principal Investigator — University of Eastern Piedmont

IPD SHARING:
Plan to Share IPD: Yes
IPD will made available for other researchers under specific request, specifying the aim. Data will be generally provided as aggregated. In case of common scientific framework, data will be provided as individual.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: as soon as databases will be ready and statistical analyses will be initiated
Access Criteria: specific request to principal investigator

REFERENCES:
- [Result] Faggiano F, Richardson C, Bohrn K, Galanti MR; EU-Dap Study Group. A cluster randomized controlled trial of school-based prevention of tobacco, alcohol and drug use: the EU-Dap design and study population. Prev Med. 2007 Feb;44(2):170-3. doi: 10.1016/j.ypmed.2006.09.010. Epub 2006 Nov 3. PMID 17084887
- [Result] Faggiano F, Galanti MR, Bohrn K, Burkhart G, Vigna-Taglianti F, Cuomo L, Fabiani L, Panella M, Perez T, Siliquini R, van der Kreeft P, Vassara M, Wiborg G; EU-Dap Study Group. The effectiveness of a school-based substance abuse prevention program: EU-Dap cluster randomised controlled trial. Prev Med. 2008 Nov;47(5):537-43. doi: 10.1016/j.ypmed.2008.06.018. Epub 2008 Jul 9. PMID 18657569
- [Result] Faggiano F, Vigna-Taglianti F, Burkhart G, Bohrn K, Cuomo L, Gregori D, Panella M, Scatigna M, Siliquini R, Varona L, van der Kreeft P, Vassara M, Wiborg G, Galanti MR; EU-Dap Study Group. The effectiveness of a school-based substance abuse prevention program: 18-month follow-up of the EU-Dap cluster randomized controlled trial. Drug Alcohol Depend. 2010 Apr 1;108(1-2):56-64. doi: 10.1016/j.drugalcdep.2009.11.018. Epub 2010 Jan 18. PMID 20080363
- [Result] Gabrhelik R, Duncan A, Miovsky M, Furr-Holden CD, Stastna L, Jurystova L. "Unplugged": a school-based randomized control trial to prevent and reduce adolescent substance use in the Czech Republic. Drug Alcohol Depend. 2012 Jul 1;124(1-2):79-87. doi: 10.1016/j.drugalcdep.2011.12.010. Epub 2012 Jan 21. PMID 22266087
- [Result] Sanchez ZM, Valente JY, Galvao PP, Gubert FA, Melo MHS, Caetano SC, Mari JJ, Cogo-Moreira H. A cluster randomized controlled trial evaluating the effectiveness of the school-based drug prevention program #Tamojunto2.0. Addiction. 2021 Jun;116(6):1580-1592. doi: 10.1111/add.15358. Epub 2021 Jan 28. PMID 33245788
- [Result] Vigna-Taglianti F, Mehanovic E, Alesina M, Damjanovic L, Ibanga A, Pwajok J, Prichard G, van der Kreeft P, Virk HK; Unplugged Nigeria Coordination Group. Effects of the "Unplugged" school-based substance use prevention program in Nigeria: A cluster randomized controlled trial. Drug Alcohol Depend. 2021 Nov 1;228:108966. doi: 10.1016/j.drugalcdep.2021.108966. Epub 2021 Aug 28. PMID 34509736
- [Result] Foxcroft DR, Tsertsvadze A. Universal school-based prevention programs for alcohol misuse in young people. Cochrane Database Syst Rev. 2011 May 11;(5):CD009113. doi: 10.1002/14651858.CD009113. PMID 21563171
- [Result] Catalano RF, Fagan AA, Gavin LE, Greenberg MT, Irwin CE Jr, Ross DA, Shek DT. Worldwide application of prevention science in adolescent health. Lancet. 2012 Apr 28;379(9826):1653-64. doi: 10.1016/S0140-6736(12)60238-4. Epub 2012 Apr 25. PMID 22538180
- [Result] Wiebe JM, Cox BJ, Mehmel BG. The South Oaks Gambling Screen Revised for Adolescents (SOGS-RA): further psychometric findings from a community sample. J Gambl Stud. 2000 Autumn;16(2-3):275-88. doi: 10.1023/a:1009489132628. PMID 14634316
- [Derived] Vigna-Taglianti FD, Martorana M, Viola E, Renna M, Vadrucci S, Sciutto A, Andra C, Mehanovic E, Ginechesi M, Vullo C, Ceccano A, Casella P, Faggiano F; GAPUnplugged Coordination Group. Evaluation of Effectiveness of the Unplugged Program on Gambling Behaviours among Adolescents: Study Protocol of the Experimental Controlled Study "GAPUnplugged". J Prev (2022). 2024 Jun;45(3):405-429. doi: 10.1007/s10935-024-00772-4. Epub 2024 Feb 28. PMID 38416313
- See also: website including information on Unplugged program, evaluation study and effectiveness — http://www.eudap.net
- See also: page of EMCDDA website describing the effectiveness of Unplugged — http://www.emcdda.europa.eu/best-practice/xchange/unplugged_en